CLINICAL TRIAL: NCT02694484
Title: Search Cytomegalovirus (CMV) in Healthy Volunteers Stools Samples Selected as Potential Donor for Fecal Microbiota Transplant
Brief Title: Search Cytomegalovirus in Healthy Volunteers Stools Samples Selected as Potential Donor for Fecal Microbiota Transplant
Acronym: TRANSFECMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: I15033 TRANSFECMV
Record Dates: First submitted 2015-12-07; First posted 2016-02-29 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: CMV; Healthy Volunteers
Keywords: Cytomegalovirus; Stool sample; Healthy Volunteers; Fecal microbiota transplant
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Other): For healthy volunteers corresponding to the inclusion criteria it will be taken them Blood and stool samples : a blood sample during the inclusion visit and if they are seropositive for the CMV, it will be taken them another blood sample and they will give a stool sample for the following visit
  Interventions: Other: Blood and stool samples

INTERVENTIONS:
Other: Blood and stool samples — Blood sample at Day 1 and blood and stool sample at the next visit

SUMMARY:
Fecal microbiota transplantation (FMT) is recommended in the treatment of recurrent Clostridium difficile infection (CDI). The principle is to administer a fecal suspension of a healthy subject (donor) in the digestive tract of a patient with an CDI (receiver). Donors are being clinical and laboratory screening to reduce the likelihood of pathogens transmission (infectious and other). Cytomegalovirus (CMV) is part of the examinations requested by the Agence national de sécurité du médicament et des produits de santé in the context of clinical research. A sero-matching between donor and recipient CMV is requested. This recommendation eliminates many potential donors to a recipient. To date, the frequency detection level of CMV in stool in healthy volunteers with documented positive CMV serology is not known. In addition, CMV transmission risk via the stool is not established. This study aims to determine the detection frequency of CMV in healthy volunteers stool samples selected as potential donors for a FMT and having a positive CMV serology documented

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 and under 65 years
* Having a normal transit (less than three stools per day and more than three bowel movements per week)
* Body mass index (BMI) <30 and> 16.9
* Accept the constraints of the study, ie two visits (inclusion and Following Visit), a stool sample, two blood tests
* Having given and signed informed consent
* Being affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Taking a treatment with anti-CMV action in three months by acyclovir, valacyclovir, ganciclovir, valganciclovir, foscarnet, cidofovir, brincidofovir
* Having an absolute exclusion criteria to donation defined by the survey of French Group Fecal Transplant:
* Digestive disorders (acute or chronic diarrhea) in the three months prior to donation
* Known chronic disease (except hypertension and hypercholesterolemia)
* Documented history of typhoid fever
* Taking long-term medication (except contraceptives, cholesterol-lowering and antihypertensive treatment)
* Antibiotic taken within three months
* Stay in tropics during the three months prior to donation,
* Residence of several years in tropics (over 24 months)
* Hospitalization abroad of more than 24 hours in the last 12 months to the donor or his entourage (those living under the same roof)
* Healthy Volunteers who have not reached the limit of compensation by social security or exclusion period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Detection frequency of CMV | 30 days
  Detection frequency of CMV in healthy volunteers stool samples with the selection criteria for the gift of fecal microbiota and having a CMV positive serology

SECONDARY OUTCOMES:
Presence of CMV in the stool and in blood. | At day 30
  Evaluation of the link between the presence of CMV in the stool and the detection of CMV viral load in whole blood.
Infectivity of CMV present in faecal | At day 30
  Evaluation of the infectivity of CMV present in faecal

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre de biologie pathologie / Laboratoire de virologie, Lille
  - Cic 1403-Crb Inserm-Chu, Lille
  - Service des Maladies Infectieuses, Lille
  - Cic - Inserm - 1435, Limoges
  - Service de Bactériologie-Virologie-Hygiène/CNR des Cytomégalovirus, Limoges

REFERENCES:
- [Result] Galperine T, Engelmann I, Hantz S, Postil D, Dewilde A, Deplanque D, Martin R, Labreuche J, Lazrek M, Somers S, Ribot E, Alain S. Cytomegalovirus in donors for fecal microbiota transplantation, the phantom menace? PLoS One. 2023 Jun 29;18(6):e0287847. doi: 10.1371/journal.pone.0287847. eCollection 2023. PMID 37384665